CLINICAL TRIAL: NCT01293175
Title: Whole Grain Polyphenol Bioavailability and Effects on Inflammatory, Oxidative and Hormonal Status
Brief Title: Whole Grain Polyphenol Bioavailability and Effects on Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Paola Vitaglione, Dr, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DSA-FF-002
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2013-07-12 (Estimated); Status verified 2013-07

CONDITIONS: Overweight
Keywords: whole grains; polyphenols; overweight; bioavailability; antioxidant status; inflammation
MeSH Terms: conditions — Overweight; Inflammation | interventions — Whole Grains

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole grains (Experimental): Subjects will consume whole grains every day for two months
  Interventions: Dietary Supplement: Whole grains
- Control (No Intervention): Subjects will consume their habitual diet

INTERVENTIONS:
Dietary Supplement: Whole grains — Subjects will consume whole grains at dose of 80 g/die, for two months
  Arms: Whole grains

SUMMARY:
Whole grains (WG) contain numerous physiologically bioactive compounds, a key group being polyphenolic compounds such as ferulic acid (FA). These whole grain polyphenolic compounds have been shown to have potent antioxidant activity. This study will evaluate bioavailability of WG bioactive compounds and their physiological impact on health outcomes, mainly related to inflammatory, oxidative and hormonal status, in overweight subjects.

DETAILED DESCRIPTION:
Epidemiological evidence indicates that consumption of whole grains (WG) is associated with improved health and decreased risk for common chronic diseases. However there is paucity of intervention data regarding the beneficial effects of WG in vascular health and associated metabolic disorders.

From 2007 up to now five main intervention studies using WG were published. The results from these studies consistently showed no efficacy of WG to modify biochemical parameters in free-living subjects including WG in their habitual diet. Anyway some drawbacks could be found and mainly regarding subject compliance to the treatment and the type of WG-rich foods supplied.

Our working hypothesis is based on WG physiologically bioactive compounds mainly polyphenolic compounds such as ferulic acid (FA). FA is covalently bound to arabinoxylans constituting WG dietary fiber. This structure represents a natural way to carry polyphenol compounds, into the lower gut. A previous work indicated that intestinal microflora particularly Bifidobacteria and Lactobacilli is able to ferment WG polysaccharide moiety (prebiotic effect) and at the same time microbial esterases can release free phenolic acids. The free acids are adsorbed through the colon barrier into the blood. The slow and continuous release of phenolic acids, particularly FA, determines an increase of baseline level of FA in the blood of WG consumers. However no study correlated FA plasma concentration with health parameters such as biomarkers of inflammation, glucose metabolism and oxidative status which may be in turn associated to the CVD risk.

In this framework a controlled, parallel, two arm intervention study will be performed using a WG-rich product that will be selected from those commercially available for having a high content of FA (>500 mg/kg). The aim of this study is to evaluate the bioavailability of FA over a two month-treatment in overweight subjects and to correlate variation of FA plasma concentrations with biomarkers of oxidative (plasma antioxidant capacity, MDA) and inflammatory (CRP, anti- and pro-inflammatory cytokines) status, with nutritional status and with gastro-intestinal hormones related to appetite and glucose metabolism (ghrelin, PYY, PP, insulin, GLP-1, GIP and leptin). Eighty subjects will be selected in the respect of strict inclusion and exclusion criteria and will be randomized to include WG in opportunely revised individual habitual diet, or to continue with their habitual diet. At baseline, after 1 month and after 2 months from starting the protocol, blood drawings will be performed and urine and feces will be collected from fasting subjects. Gastro-intestinal hormone response and glucose metabolism following a standard meal will be also evaluated at baseline and at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 years old, male and female
* Healthy by medical assessment
* Overweight: BMI > 25 and < 32 kg/m2
* Habitual diet characterized by i) absence of WG (all dietary carbohydrates derived from refined cereals); ii) absence of pro-biotics; iii) intake of dietary fibre ≤ 10 g/d; iv) intake of fruit and vegetables ≤ 2 portions/die; v)habit to have breakfast
* Sign of a written informed consent

Exclusion Criteria:

* Age < 18 and > 60 years old
* Pregnancy or breastfeeding
* Fasting plasma triglycerides ≥ 200 mg/dl and cholesterol > 200 mg/dl
* Cardiovascular events (AMI and/or stroke) in the last 6 months
* Regular intensive physical activity
* Hypertension
* Intestinal or metabolic diseases/disorders such as diabetic, renal, hepatic, pancreatic or ulcer
* Previous abdominal/gastrointestinal surgery
* Regular consumption of medication
* Antibiotic therapy within 2 months previous the study
* Food allergies and intolerances (celiac disease, lactose intolerance,)
* Concurrent participation or having participated in another clinical trial during the last 3 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Variation of serum polyphenol concentration | 1 year
  Measure of serum polyphenol concentration (nmol/L)
Variation of plasma lipids | 1 year
  Measure of plasma concentrations (mg/dL) of Total-, LDL-, and HDL-Cholesterol, as well as Triglycerides

SECONDARY OUTCOMES:
Variation of serum antioxidant capacity | 1 year
  Measure of plasma FRAP (µmol/L) and MDA (µmol/L) concentrations.
Variation of body weight | 1 year
  Measure of body weight (kg)
Variation of serum inflammatory marker concentration | 1 year
  Measure of serum CRP, IL-6, TNF-α, PAI-1, Visfatin, Resistin concentration (pg/mL)
Variation of fecal microbiota composition | 1 year
  By FISH (colony-forming unit, CFU/g)
Variation of serum gastro-intestinal hormone concentration | 1 year
  It will be evaluated following a standard meal test. In particular plasma response (pg/mL) of Ghrelin, PYY, Leptin, GIP, GLP-1, PP and insulin will be assessed
Variation of blood pressure | 1 year
  Measure of blood pressure (mmHg)
Variation of body circumferences | 1 year
  Measure of waist and hip circumferences (mm)
Variation of body composition | 1 year
  Measure of body composition (% of lean and fat mass, % water)

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Fogliano, Prof, Study Director — University of Naples; Paola Vitaglione, Dr, Principal Investigator — University of Naples
Locations (1):
- Department of Food Science, Portici, Italy

REFERENCES:
- [Derived] Vitaglione P, Mennella I, Ferracane R, Rivellese AA, Giacco R, Ercolini D, Gibbons SM, La Storia A, Gilbert JA, Jonnalagadda S, Thielecke F, Gallo MA, Scalfi L, Fogliano V. Whole-grain wheat consumption reduces inflammation in a randomized controlled trial on overweight and obese subjects with unhealthy dietary and lifestyle behaviors: role of polyphenols bound to cereal dietary fiber. Am J Clin Nutr. 2015 Feb;101(2):251-61. doi: 10.3945/ajcn.114.088120. Epub 2014 Dec 3. PMID 25646321